CLINICAL TRIAL: NCT06997848
Title: The Application of Ultrasound in the Evaluation of Patients With Colon Cancer-related Obstruction Receiving Colonic Stent Placement
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Principal Investigator, National Taiwan University Hospital
Other Study IDs: 202112159RINB
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Resolution of Bowel Obstruction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: colonic stent — colonic stent deployment

SUMMARY:
Bowel ultrasound may serve as a diagnostic tool to detect the resolution of bowel obstruction. In this study, we aim to validate the use of bowel ultrasound to evaluate patients with colon obstruction receiving colonic stents at National Taiwan University Hospital from January 2010 to June 2023. We will investigate the association between decompression of the ascending colon and the following surgical procedure, complication, and occurrence of bacteremia.

ELIGIBILITY:
Inclusion Criteria: acute colorectal obstruction without perforation due to malignancy or extra-colonic tumor.

Exclusion Criteria: acute colorectal obstruction with perforation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: acute colorectal obstruction without perforation due to malignancy or extra-colonic tumor.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
the ascending colon diameter and wall thickness | 2 days
  the diameter and thickness before abd after the stent

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Ching Lien, Principal Investigator — NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan